CLINICAL TRIAL: NCT00489983
Title: A Multicenter Phase 2 Randomized Trial of Single-Agent ALIMTA or ALIMTA With Sequentially Administered GEMZAR as First-Line Chemotherapy in Elderly Patients or Patients Who Are Not Eligible for Platinum-Based Chemotherapy With Advanced NSCLC
Brief Title: Trial of Pemetrexed or Pemetrexed With Gemcitabine for Patients With Advanced Lung Cancer Who Are Not Eligible for Platinum-Based Chemotherapy and Have Not Previously Been Treated With Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5119; H3E-EW-JMEM
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: pemetrexed
Drug: gemcitabine

SUMMARY:
This study is for elderly patients who haven't been given prior chemotherapy or for patients who cannot be treated with platinum based chemotherapy. The patients who are eligible for this study will have been diagnosed with advanced or metastatic non-small cell lung cancer. The patients will be randomly assigned to one of two treatment options: single agent pemetrexed or single agent pemetrexed with single agent gemcitabine following right after the pemetrexed treatment.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed NSCLC not amenable to surgery or radiotherapy of curative intent
* locally advanced or metastatic Stage IIIb (with N3 supraclavicular or T4 for pleural effusion) or IV NSCLC
* no prior chemotherapy
* measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria (Therasse et al. 2000)
* men and women greater than or equal to 70 years of age or patients who, in the investigator's opinion, are not eligible for platinum-based chemotherapy

Exclusion Criteria:

* have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* have symptomatic brain metastases
* have a history or presence of other malignancy except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years before without recurrence (excluding melanoma, breast cancer and hypernephroma)
* are unable to interrupt therapy with aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs) such as naproxen, piroxicam, diflunisal, or nabumetone around each dose of pemetrexed (5 days for short-acting or 8 days for long acting preparations)
* are unable or unwilling to take steroids
* are unable or unwilling to take folic acid or vitamin B12 supplementation
* have clinically detectable (by physical examination) third-space fluid collections; for example, ascites or pleural effusions that cannot be controlled by drainage or other procedures prior to study entry
* have other serious concomitant illness or medical conditions according to investigator criteria, including but not limited to the following:

  * congestive heart failure or angina pectoris, except if it is medically controlled
  * previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension, or arrhythmias
  * active infection requiring iv antibiotics
  * active ulcer, unstable diabetes mellitus, or other contra-indication to corticotherapy
  * superior vena cava syndrome

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 91 (Actual)
Dates: Start 2003-07; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
To evaluate efficacy.

SECONDARY OUTCOMES:
To evaluate toxicity.
To evaluate response.
To evaluate overall survival, duration of overall response, and duration of stable disease.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin, Germany
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan, Italy
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, United Kingdom

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com